CLINICAL TRIAL: NCT01465386
Title: A Phase II Study of Subcutaneous Bortezomib as Maintenance Therapy for Patients With High-risk Acute Myeloid Leukemia in Remission
Brief Title: Bortezomib in Treating Patients With High-Risk Acute Myeloid Leukemia in Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early due to slow enrollment
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2529.00; NCI-2011-03115 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-10; First posted 2011-11-04 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive bortezomib SC on days 1, 8, 15 and 22. Treatment repeats every 35 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given SC
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial studies how well bortezomib works in treating patients with high-risk acute myeloid leukemia (AML) in remission. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if bortezomib when given as maintenance therapy for six months post-remission can improve the progression-free survival (PFS) rate by 50% (or 4.5 months) in first remission patients with high-risk AML.

SECONDARY OBJECTIVES:

I. To determine the overall survival (OS) after maintenance therapy with bortezomib in first remission AML patients.

II. To assess the safety and tolerability of subcutaneous (SC) administration of bortezomib given as maintenance therapy to first remission AML patients.

OUTLINE:

Patients receive bortezomib SC on days 1, 8, 15 and 22. Treatment repeats every 35 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, every 3 months for 2 years, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All adults with first remission AML including those with prior myelodysplasia (MDS)/AML, therapy-related AML, AML with trilineage dysplasia (AML-TLD), and AML with adverse cytogenetics
* History of histopathologically documented AML that is currently in first remission with the presence of 5% or less blasts by morphology and/or flow cytometry from a bone marrow aspirate and/or biopsy obtained within 14 days of enrollment
* Patients must start therapy between 3-8 weeks after receiving their last prior therapy (either induction therapy or consolidation therapy)
* Patients may receive up to 4 courses of remission consolidation therapy (e.g., cytarabine) prior to enrollment
* Normal kidney and liver function with serum creatinine =< 2.0 mg/dl
* Total bilirubin =< 1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Male subjects, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse
* Understand and voluntarily sign the informed consent form for this study

Exclusion Criteria:

* Favorable AML features defined as the following:

  * t(8;21)(q22;q22); RUNX1-RUNX1T1
  * inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11
  * Mutated NPM1 without FLT3-ITD (normal karyotype)
  * Mutated CEBPA (normal karyotype)
* Persistent clinically significant non-hematological toxicity that is > Grade 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4 from prior chemotherapy
* Active uncontrolled infection
* Known infection with human immunodeficiency virus (HIV)
* Medical condition, serious concurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize patient safety or interfere with the objectives of the study
* Uncontrolled or significant cardiovascular disease, including:

  * Uncontrolled angina or myocardial infarction within 6 months
  * Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, unless a screening echocardiogram (ECHO) or Multiple Gate Acquisition Scan (MUGA) performed within 1 month prior to study screening results in a left ventricular ejection fraction (LVEF) that is >= 45% (or institutional lower limit of normal value)
  * Prolonged QTc interval (> 450 msec)
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patient has a platelet count of < 30,000 within 3 days before enrollment
* Patient has an absolute neutrophil count of < 300 within 3 days before enrollment
* Patient has >= Grade 2 peripheral neuropathy
* Patient has hypersensitivity to bortezomib, boron, or mannitol
* Female patients who are lactating or have a positive urine pregnancy test during the screening; pregnancy testing is not required for postmenopausal or surgically sterilized women
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01-28 (Actual); Study Completion 2015-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Patients: Patients receive bortezomib SC on days 1, 8, 15 and 22. Treatment repeats every 35 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  bortezomib: Given SC
Period: Overall Study
Arm/Group | Treated Patients
Started | 6
Completed | 2
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 78 [61 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Number of days from enrollment to recurrence of acute myeloid leukemia as determined by the reappearance of blasts in the blood or marrow
Time Frame: Up to 2 years
Population: Patient who began maintenance treatment with bortezomib after induction of remission
Measure: Median (Full Range); unit: days
Units Other Than Participants: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 6
days | 107 [14 to 575]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=6)
Altered Mental Status (Nervous system disorders) | 1 (1) — Serious as required hospitalization, but not related to study drug
Cholechystitis (Gastrointestinal disorders) | 1 (1) — Serious as required hospitalization, but not related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=6)
Peripheral neuropathy (Nervous system disorders) | 1 (1) — Grade 2 peripheral neuropathy, a known adverse effect of study drug

LIMITATIONS AND CAVEATS:
Difficulty finding patients willing or available to come in to clinic for weekly injections for the duration of the study. Study was ultimately closed because of slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes